CLINICAL TRIAL: NCT01525914
Title: Assessment of Response of Patients on Surveillance for Favorable Risk Prostate Cancer to Dutasteride
Brief Title: Response of Patients on Surveillance for Prostate Cancer to Dutasteride
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Toronto Sunnybrook Regional Cancer Centre (Other)
Responsible Party: Principal Investigator, Dr. Laurence Klotz, Principal Investigator, Sunnybrook Health Sciences Centre
Other Study IDs: CRT114918
Record Dates: First submitted 2011-09-22; First posted 2012-02-03 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; PSA kinetics; PSA doubling time; active surveillance
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — prostate biopsy tissue stored on site
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dutasteride, active surveillance: men with favorable risk prostate cancer on surveillance treated with dutasteride
  Interventions: Drug: Dutasteride

INTERVENTIONS:
Drug: Dutasteride — dutasteride 0.5mg daily
  Other Names: Avodart

SUMMARY:
Hypothesis: That, in men on surveillance for favorable risk prostate cancer treated with dutasteride, prostate specific antigen (PSA) kinetics is of value in identifying those men who harbor occult high grade prostate cancer.

The study will determine the prevalence of a secondary rise in PSA > 0.5 ng/ml and the PSA doubling time in subjects on surveillance being treated with dutasteride.

DETAILED DESCRIPTION:
This analysis is a subset of the data associated with the active surveillance cohort at Sunnybrook Health Sciences Centre. Approximately 150 subjects within the cohort have received dutasteride therapy from 6 months to 3 years. All subjects have had serial PSAs at regular intervals between 3 to 6 months, and all have had a biopsy performed within 1 to 3 years of initiating dutasteride. The prevalence of a secondary rise in PSA > 0.5ng/ml will be calculated with the impact of dutasteride therapy on the PSA doubling time. This information will be correlated with baseline PSA value, prostate volume, extent of disease on initial biopsy and baseline PSA kinetics. PSA kinetics will be also correlated with Gleason score upgrading on repeat biopsy. The rate of negative biopsies in men on dutasteride therapy will be compared with a similar group of surveillance subjects not treated with dutasteride.

ELIGIBILITY:
Inclusion Criteria:

* Patients on active surveillance for favorable risk prostate cancer who have been treated with dutasteride following the diagnosis of cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are a subset of the men with prostate cancer on surveillance for favorable risk prostate cancer cohort
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
change in serum PSA | change from baseline in serum PSA up to secondary rise in serum PSA > 0.5, up to 6 months
  The time that the change in serum PSA from baseline to the secondary rise will be used to determine the PSA 'kinetics' in men on surveillance for prostate cancer.

SECONDARY OUTCOMES:
rate of secondary rise in serum PSA | at 6 months after starting dutasteride therapy
  Rate of rise in sereum PSA will be correlated with prostate gland volume at initial biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Klotz, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada